CLINICAL TRIAL: NCT07354737
Title: Efficacy and Safety of a Voltage-Guided Stepwise Strategy for Pulmonary Vein Isolation: A Randomized Comparison With Conventional Circumferential Antral Pulmonary Vein Isolation
Brief Title: Efficacy and Safety of a Voltage-Guided Stepwise Strategy for Pulmonary Vein Isolation
Acronym: VoS-PVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Kwang-No Lee, Associate Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AJIRB-MED-INT-20-475
Record Dates: First submitted 2026-01-18; First posted 2026-01-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF); Atrial Fibrillation Ablation Procedure; Atrial Tachyarrhythmia Recurrence; Esophageal Thermal Injury
Keywords: Atrial fibrillation; Catheter ablation; Pulmonary vein isolation; Voltage-guided ablation; High-density voltage mapping; Segmental ablation; Randomized controlled trial; Noninferiority trial
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1 to one of two pulmonary vein isolation strategies (voltage-guided stepwise PVI vs conventional circumferential antral PVI) and followed in parallel for 12-month atrial tachyarrhythmia recurrence and safety outcomes.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are masked to treatment assignment. Treating physicians/operators are not masked due to the nature of the catheter ablation strategies. Atrial tachyarrhythmia recurrence is assessed using scheduled ECG and ambulatory monitoring and reviewed by treating clinicians who are aware of group allocation. Outcomes assessors for safety endpoints are masked to treatment assignment for evaluation of post-procedure endoscopic findings using prespecified criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Voltage-guided Stepwise Pulmonary Vein Isolation (PVI) (Experimental): Participants undergo catheter ablation for atrial fibrillation using a voltage-guided stepwise PVI strategy. Ablation is delivered point-by-point along a predefined antral line, starting in higher-voltage regions and expanding stepwise to lower-voltage regions only as needed until pulmonary vein isolation is achieved. Additional ablation may be performed if required to complete isolation based on residual electrical signals.
  Interventions: Device: Radiofrequency ablation catheter system
- Conventional Circumferential Antral Pulmonary Vein Isolation (PVI) (Active Comparator): Participants undergo catheter ablation for atrial fibrillation using a conventional circumferential antral PVI strategy. A continuous circumferential lesion set is created around the pulmonary vein antrum to achieve isolation. Additional ablation may be performed if required to complete isolation based on residual electrical signals.
  Interventions: Device: Radiofrequency ablation catheter system

INTERVENTIONS:
Device: Radiofrequency ablation catheter system — Catheter ablation for atrial fibrillation performed using a voltage-guided stepwise PVI strategy. Ablation is delivered point-by-point along a predefined antral line, starting at higher-voltage sites and expanding stepwise to lower-voltage sites only as needed until pulmonary vein isolation is achieved. Additional potential-guided ablation may be performed if required to complete isolation.
  Other Names: Voltage-guided stepwise PVI
  Arms: Voltage-guided Stepwise Pulmonary Vein Isolation (PVI)
Device: Radiofrequency ablation catheter system — Catheter ablation for atrial fibrillation performed using a conventional circumferential antral PVI strategy. A continuous circumferential lesion set is created around the pulmonary vein antrum to achieve isolation. Additional potential-guided ablation may be performed if required to complete isolation.
  Other Names: Conventional circumferential antral PVI
  Arms: Conventional Circumferential Antral Pulmonary Vein Isolation (PVI)

SUMMARY:
The goal of this clinical trial is to learn if a voltage-guided stepwise pulmonary vein isolation (PVI) strategy can achieve effective PVI while potentially reducing lesion delivery, compared with conventional circumferential antral PVI, in adults (≥20 years) with paroxysmal or non-paroxysmal atrial fibrillation undergoing first-time catheter ablation. The main question(s) it aims to answer is/are:

Is voltage-guided stepwise PVI non-inferior to conventional circumferential antral PVI for atrial tachyarrhythmia recurrence within 12 months after ablation?

Does voltage-guided stepwise PVI differ from conventional circumferential antral PVI in procedural characteristics and safety outcomes, including endoscopically detected esophageal thermal injury and acute procedural complications?

Researchers will compare the voltage-guided stepwise PVI arm to the conventional circumferential antral PVI arm to see if the stepwise approach maintains arrhythmia outcomes while changing lesion delivery requirements and safety outcomes.

Participants will:

Be randomized 1:1 to undergo catheter ablation with either voltage-guided stepwise PVI or conventional circumferential antral PVI.

Undergo diagnostic esophagoscopy between post-procedure day 1 and day 3 to systematically assess for esophageal thermal injury.

Complete follow-up evaluations at 3, 6, 9, and 12 months (and every 6 months thereafter), including 12-lead ECGs and 24- or 72-hour Holter monitoring.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) catheter ablation is commonly performed using pulmonary vein isolation (PVI). Conventional PVI is achieved by creating a continuous circumferential antral lesion set, but this may require extensive lesion delivery on the posterior left atrium where the esophagus is adjacent. Voltage mapping can characterize regional atrial signal amplitude, and a stepwise strategy that prioritizes higher-voltage sites along a planned antral path may reduce unnecessary lesion delivery while still achieving acute isolation. This randomized trial compares a voltage-guided stepwise PVI strategy with a conventional circumferential antral PVI strategy in patients undergoing first-time AF ablation.

Participants are randomized 1:1 to one of two PVI strategies. All procedures are performed using a standardized workflow for left atrial mapping and PVI verification. Acute PVI is confirmed by elimination or dissociation of pulmonary vein potentials. Durability of isolation is assessed during the index procedure using adenosine testing for dormant conduction, and trigger provocation is performed per protocol. If isolation is incomplete, additional ablation guided by residual electrical potentials is permitted in both groups to achieve the procedural endpoint.

In the voltage-guided stepwise PVI group, ablation is delivered point-by-point along a predefined antral line using a prespecified stepwise algorithm. Lesion delivery is initiated at sites meeting a high bipolar voltage threshold and expanded stepwise to include progressively lower-voltage sites only as needed until PVI is achieved. If isolation cannot be achieved at the minimum voltage threshold, previously ablated points may be connected to complete a continuous line, and adjunctive ablation (e.g., carina or residual potential-guided ablation) may be performed when necessary.

In the conventional circumferential antral PVI group, operators create a continuous circumferential antral lesion set around the pulmonary veins using the standard approach. Additional potential-guided ablation is allowed when needed to achieve PVI. Voltage information is not used to guide lesion distribution in this group during the procedure.

To systematically assess esophageal safety, diagnostic esophagoscopy is performed between post-procedure day 1 and day 3 in all participants using prespecified criteria for esophageal thermal injury. Follow-up is conducted at scheduled intervals with electrocardiography and ambulatory rhythm monitoring per protocol to document arrhythmia outcomes. A post-ablation blanking period is applied for clinical outcome assessment.

Analyses are performed primarily on an intention-to-treat basis. In addition to the prespecified efficacy and safety comparisons between treatment groups, exploratory analyses evaluate relationships between local voltage characteristics and the voltage threshold required for isolation, including variation by pulmonary vein location and AF phenotype.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years
* Symptomatic paroxysmal or non-paroxysmal atrial fibrillation
* Scheduled for first-time catheter ablation with pulmonary vein isolation
* Able to provide written informed consent

Exclusion Criteria:

* Prior catheter or surgical ablation for atrial arrhythmia
* Myocardial infarction within the past 3 months
* Stroke or transient ischemic attack within the past 6 months
* New York Heart Association (NYHA) class III-IV heart failure
* Contraindication to oral anticoagulation
* Pregnancy
* Any medical condition judged by the investigator to make participation unsafe or to interfere with study procedures or follow-up

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
Atrial tachyarrhythmia recurrence within 12 months after the index ablation | 12 months after the index ablation (excluding a 3-month blanking period)
  Recurrence of atrial tachyarrhythmia (atrial fibrillation, atrial flutter, or atrial tachycardia) within 12 months after the index ablation, defined as an episode documented on a 12-lead ECG or lasting ≥30 seconds on ambulatory monitoring (24-72-hour Holter). Events occurring during the 3-month post-ablation blanking period are excluded.

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-No Lee, MD, PhD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University Hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in publications from this trial, along with the data dictionary, will be made available to qualified researchers upon reasonable request. Requests must include a brief research proposal and analysis plan and will be reviewed by the study team for scientific merit, feasibility, and protection of participant privacy. Access will require execution of a data use agreement and, when applicable, institutional ethics approval. Shared data will be limited to the minimum necessary and will exclude direct identifiers; recipients must agree not to attempt re-identification or onward sharing without permission.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication of the primary results and ending 5 years thereafter.
Access Criteria: Access to de-identified IPD will be provided to qualified researchers upon reasonable request. Requestors must submit a brief research proposal, analysis plan, and evidence of relevant qualifications. Requests will be reviewed by the study team for scientific merit, feasibility, and protection of participant privacy. Access will be granted after execution of a data use agreement and confirmation of institutional ethics approval where required. Data will be shared via a secure method, limited to the minimum necessary dataset, and recipients must agree not to attempt re-identification or share the data with third parties without written permission.